CLINICAL TRIAL: NCT05414721
Title: The Effects of Low Flow and Normal Flow Desflurane Anesthesia on Postoperative Liver and Renal Functions and Serum Cystatin C Levels in Geriatric Patients: A Prospective Randomized Controlled Study
Brief Title: The Effects of Low Flow and Normal Flow Desflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacı Yusuf Güneş, Assistant proffesor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/05-07
Record Dates: First submitted 2022-05-24; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia; Liver Functions; Kidney Functions; Geriatric
Keywords: Low flow desflurane anesthesia,; Liver functions; Kidney functions; Serum cystatin C levels; Geriatric patients.

STUDY DESIGN:
Intervention Model Description: Sixty patients were included in the study. The patients were randomly divided into two groups as low flow anesthesia and normal flow anesthesia. All patients were preoxygenated. Midazolam, fentanyl, propofol and rocuronium were administered iv for induction of anesthesia. After intubation all patients were mechanically ventilated with 50%O2+50% air+7% desflurane in a 4L/min fresh gas flow until the MAC value reached to 1.
  When the MAC value of desflurane was 1, the fresh gas flow was reduced to 0.5L/min (60%O2+40%air) in GroupD.
  In GroupN, the fresh gas flow was reduced to 2L/min (40%O2+60% air). The anesthesia was maintained in these fresh gas flows. HR, SBP, DBP, MBP, SpO2 and BIS values were recorded preanesthesia and during surgery. To research the liver and the kidney functions, blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low flow desflurane anesthesia (Group D) (Active Comparator): All patients were preoxygenated for three minutes. Midazolam 0.03 mg/kg, fentanyl 1.5 mcg/kg , propofol 2 mg/kg and rocuronium 0.6 mg/kg were administered iv for induction of anesthesia. After intubation all patients were mechanically ventilated with 50% O2+50% air + 6-7% desflurane in a 4 L/min fresh gas flow until the MAC value reached 1. When the MAC value of desflurane was 1, fresh gas flow was decreased to 0.5 L/min (60% O2+40% air) in Group D. Hemodynamic parameters, SpO2 and BIS values were recorded after induction, at the beginning of low flow/normal flow anesthesia and every 5 minutes during surgery. The patients were observed in terms of side effects and complications during the operation and in the postoperative period. To research the liver and the kidney functions, blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
  Interventions: Drug: Low flow desflurane anesthesia (Group D)
- Normal flow desflurane anesthesia (Group N) (No Intervention): All patients were preoxygenated for three minutes. Midazolam 0.03 mg/kg, fentanyl 1.5 mcg/kg , propofol 2 mg/kg and rocuronium 0.6 mg/kg were administered iv for induction of anesthesia. After intubation all patients were mechanically ventilated with 50% O2+50% air + 6-7% desflurane in a 4 L/min fresh gas flow until the MAC value reached 1. When the MAC value of desflurane was 1, fresh gas flow was decreased to 2 L/min (40% O2+60% air) in Group N. Hemodynamic parameters, SpO2 and BIS values were recorded after induction, at the beginning of low flow/normal flow anesthesia and every 5 minutes during surgery. The patients were observed in terms of side effects and complications during the operation and in the postoperative period. To research the liver and the kidney functions, blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.

INTERVENTIONS:
Drug: Low flow desflurane anesthesia (Group D) — When the MAC value of desflurane was 1, fresh gas flow was decreased to 0.5 L/min (60% O2+40% air). Hemodynamic parameters, SpO2 and BIS values were recorded after induction, at the beginning of low flow/normal flow anesthesia and every 5 minutes during surgery. The patients were observed in terms of side effects and complications during the operation and in the postoperative period. To research the liver and the kidney functions, blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
  Other Names: Normal flow desflurane anesthesia (Group N)
  Arms: Low flow desflurane anesthesia (Group D)

SUMMARY:
Aging is a physiological process. In the elderly, loss of functional reserve in all organ system, regression in anabolic processes and increase in catabolic processes are observed s (1). The number of geriatric patients is also increasing in our country. Technological developments in anesthesia and surgery technics show that we will provide medical services to more elderly patients over time(2). Cystatin C is excreted only by the kidney (7, 8). Serum cystatin C level is not affected by body muscle mass, age and gender. The half-life is short. Because of all these features, it is thought to be more sensitive than creatinine in evaluating kidney functions (8,9). In this study, it was aimed to compare the effects of low flow and normal flow desflurane anesthesia applied in geriatric patients on postoperative liver and kidney functions and serum cystatin C levels.

DETAILED DESCRIPTION:
This prospective, randomized-controlled, observational study was approved by the ethics committee of Van Yuzuncu Yıl University (Date: 16.04.2021, Decision no: 05-27). The study was performed according to the World Medical Association's Declaration of Helsinki. All enrolled patients provided written informed consent.

In this prospective study; the patients were randomly divided into 2 groups according to the fresh gas flow applied. 'Group D' (n=30) was given to the low flow anesthesia group; the group in which normal flow anesthesia was administered was named 'Group N' (n=30).

Before anesthesia, automatic calibration of the anesthesia device (Primus, Drager) and leak tests were performed. In addition, the leak test was repeated manually for each patient. Alarm limits of the anesthesia device; The lower limit of inspired oxygen concentration (FiO2) was set to 30%, upper limit of inspired CO2 to 3%, and upper limit of end-tidal carbon dioxide (etCO2) to 45 mmHg.

The disconnection alarm was set to be 5 cmH2O lower than the peak pressure, the occlusion alarm was set to 30 cmH2O, the lower expiratory gas volume lower limit was set to be 500 mL below the desired minute volume (MV).

Soda lime (Sorbo-lime, Berkim, Turkey) was used as carbon dioxide absorbent. Soda lime was checked frequently for color and changed at appropriate times. Disposable anesthesia circuit and bacterial filter were used for each case.

Electrocardiography (ECG), peak heart rate (CTA), peripheral oxygen saturation (SpO2), non-invasive blood pressure and bispectral index (BIS) monitorisation (A-2000 Aspect medical systems, USA) were performed on all patien.

As a standard, vascular access was established with a 20-gauge (G) intraket from the dorsal of the hand or antecubital fossa in each patient and, a balanced electrolyte solution was infused of 8-10 ml/kg/hr.

All patients were preoxygenated with 100% O₂ for three minutes. For anesthesia induction, 0.03 mg/kg midazolam, 1-1.5 mcg/kg fentanyl, 2 mg/kg propofol and 0.6 mg/kg rocuronium were administered iv. Intubation was performed after adequate muscle relaxation was achieved. During mechanical ventilation; Tidal volume, PEEP, respiratory rate, etCO₂, and inspiration:expiration ratio were adjusted to be 7-10 ml/kg, 5 cmH2O, 12-14/min, 30-40 mmHg, 1:2 respectively.

Both groups were given a mixture of 50% O2 + 50% air + 6-7% desflurane in a 4 L/min fresh gas flow (FGF) until the minimum alveolar concentration (MAC) value was 1.

When the MAC value of desflurane was 1, FGF was reduced to 0.5 L/min (60% O2+40% dry air+8% desflurane) in Group D. In Group N, anesthesia was maintained by reducing FGF to 2 liters per minute (40% O2+60% air+6% desflurane). It was aimed to keep the MAC value between 0.9-1.1 and BIS values between 40-60 by titration of desflurane in all patients. Hemodynamic data, SpO2 and BIS values of the patients were recorded. It was recorded before induction, after induction, when switching to low/normal flow anesthesia, and during extubation.

Venous blood samples were obtained before induction, after surgery, and at the postoperative 24th hour to evaluate liver and kidney functions.

The SPSS 27.0 program was used to evaluate the data obtained in this study. In the descriptive statistics of the data, mean, standard deviation, median minimum, maximum, frequency and ratio values were used. The distribution of variables was measured with the Kolmogorov-Smirnov test. The mann-whitney u test was used in the analysis of quantitative independent data. Wilcoxon test was used in the analysis of dependent quantitative data. Chi-square test was used in the analysis of qualitative independent data, and the fischer test was used when the chi-square test conditions were not met. Statistical significance value was accepted as p<0.05 in all tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) status of class I-III,
* Aged between 65 and 100 years,
* Scheduled to undergo general anesthesia and, the surgeries that will take longer than 1 hour.

Exclusion Criteria:

* ASA class ≥ III patients
* Thorasic surgery
* Neurosurgery
* Cardiorespiratory disease,
* Uncontrolled diabetes mellitus,
* Coagulation disorders,
* Preoperative liver and renal dysfunction,
* History of malignant hyperthermia,
* Using nephrotoxic or hepatotoxic drugs,
* Major bleeding (>1000 cc) is predicted in the operation,
* Chronic alcoholism,
* Patients with drug use or withdrawal symptoms

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Alanin Aminotransferaz (ALT) | 24 hours
  To research the serum alanin Aminotransferaz (ALT) , blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
Aspartat Aminotransferaz (AST) | 24 hours
  To research the serum Aspartat Aminotransferaz (AST) , blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
Serum creatinine | 24 hours
  To research the serum creatinine , blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
Serum cystatin C | 24 hours
  To research the Serum cystatin C , blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.
Blood urea nitrogen (BUN) | 24 hours
  To research the Blood urea nitrogen (BUN) , blood samples were taken pre-induction, post-surgery, and at the postoperative 24th hour by venous route.

SECONDARY OUTCOMES:
Heart rate (HR) | 6 hours
  HR were recorded before anesthesia induction and during surgery.
Systolic blood pressure (SBP) | 6 hours
  SBP were recorded before anesthesia induction and during surgery.
Diastolic blood pressure (DBP) | 6 hours
  DBP were recorded before anesthesia induction and during surgery.
Mean blood pressure (MBP) | 6 hours
  MBP were recorded before anesthesia induction and during surgery.
Drug allergies | 24 hours
  The patients were observed in terms of drug allergies, during the operation and in the postoperative period.
Nausea-vomiting | 24 hours
  The patients were observed in terms of nausea-vomiting during the operation and in the postoperative period.
Shivering and agitation | 24 hours
  The patients were observed in terms of shivering and agitation during the operation and in the postoperative period.
İnsufficient depth of anesthesia | During surgery
  The patients were monitored with BİS monitorization for complications such as nsufficient depth of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hacı Yusuf YG Güneş, Assist.prof, Principal Investigator — Van Yüzüncü Yıl University Van, Turkey
Locations (1):
- Van Yüzüncü Yıl University, Faculty of Medicine, Van, Tusba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be share for other resarchers.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months
Access Criteria: The access can be provided via the e-mail addresses below hyusufgunes@hotmail.com

REFERENCES:
- [Background] Horwitz M, Jakobsson JG. Desflurane and sevoflurane use during low- and minimal-flow anesthesia at fixed vaporizer settings. Minerva Anestesiol. 2016 Feb;82(2):180-5. Epub 2015 Jul 22. PMID 26198766
- [Background] Xie G, Jiang H. Clinical study of desflurane on low flow anesthesia compared with sevoflurane and enflurane. Chin Med J (Engl). 1997 Sep;110(9):707-10. PMID 9642331
- [Background] Baum JA, Aitkenhead AR. Low-flow anaesthesia. Anaesthesia. 1995 Oct;50 Suppl:37-44. doi: 10.1111/j.1365-2044.1995.tb06189.x. PMID 7485917